CLINICAL TRIAL: NCT01258075
Title: Colesevelam Oral Suspension as Monotherapy or Add-on to Metformin Therapy in Pediatric Subjects With Type 2 Diabetes Mellitus
Brief Title: Colesevelam for Children With Type 2 Diabetes
Acronym: WELKid DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEL-A-U307
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Blood glucose; Anti-diabetic; Bile acid sequestrant; Colesevelam HCl; Oral suspension; Pediatric; Add-on therapy; Add-on to metformin; Metformin; Adolescent; Lipid
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Colesevelam (Experimental): High-dose colesevelam suspended in a drink for oral administration once daily with dinner
  Interventions: Drug: High-dose colesevelam
- Placebo proxy (Experimental): Low-dose colesevelam suspended in a drink for oral administration once daily with dinner
  Interventions: Drug: Low-dose colesevelam

INTERVENTIONS:
Drug: High-dose colesevelam — 3.75 grams colesevelam hydrochloride in oral suspension
  Other Names: Welchol oral suspension
  Arms: Colesevelam
Drug: Low-dose colesevelam — 0.625 grams colesevelam hydrochloride in oral suspension
  Other Names: Welchol oral suspension
  Arms: Placebo proxy

SUMMARY:
This study will evaluate the efficacy and safety of the study drug in treating type 2 diabetes in children 10 to 17 years old.

The groups will be low-dose (0.625 g Welchol) and high-dose (3.75 g Welchol). The children will have a 2 in 5 chance of being assigned to the low-dose group. They will have a 3 in 5 chance of being assigned to the high-dose group.

We believe the study drug will be safe, well tolerated, and improve blood sugar control in children 10 to 17 years old.

DETAILED DESCRIPTION:
Colesevelam oral suspension will be studied as treatment of type 2 diabetes mellitus (T2DM) to evaluate clinical safety and efficacy in patients aged 10-17 years. The patients may have been treated with Metformin or have had no antidiabetic drug treatment in the previous three months.

Study Hypothesis: Colesevelam oral suspension for pediatric subjects with T2DM is safe, well tolerated, and shows improved blood sugar control (as evidenced by a significant change from baseline in hemoglobin A1C [HbA1c]).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus, as defined by the American Diabetes Association;
* Written informed consent of study participation
* Males and females aged 10 to 17 years, inclusive, at randomization (randomization must occur before 18th birthday);
* HbA1c at screening between 7.0% and 10.0%, inclusive;
* Fasting C-peptide >0.6 ng/mL; and
* Anti-diabetic treatment at screening:

  * Treatment-naïve or untreated; OR
  * On metformin monotherapy: Metformin monotherapy has been initiated prior to screening.

Exclusion Criteria:

* Fasting plasma glucose >270 mg/dL;
* Diagnosis of type 1 diabetes;
* History of more than one episode of ketoacidosis after the initial diagnosis of type 2 diabetes mellitus;
* Clinical laboratory assessments/evaluations, eg. autoimmune markers, aminotransferases, triglycerides, creatinine clearance, and Hb variants, that are not within the protocol-defined parameters
* Systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥95 mmHg
* Use of medications not allowed by protocol-defined parameters, eg. insulin or any medication that affects insulin sensitivity or secretion, growth hormones/somatotropin, or anabolic steroids
* Genetic syndrome or disorder known to affect glucose
* Participation in a weight loss program or another interventional research study within 60 days;
* Female participants who are lactating, pregnant, or plan to become pregnant within 1 year of screening;
* Female participants who are sexually active and unwilling to use appropriate contraception for the duration of the study;
* History of bowel obstruction;
* Other significant organ system illness or condition (including psychiatric or developmental disorder) that, in the opinion of the Investigator, would prevent full participation

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2011-02-24 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader/Medical Monitor, Study Director — Daiichi Sankyo
Locations (23):
- United States (23):
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - Oakland, California
  - San Diego, California
  - Aurora, Colorado
  - Hartford, Connecticut
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - New York, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- See also: product information, FDA-approved labeling, usage instructions, dosage forms available — http://www.welchol.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 236 participants who met all inclusion criteria and no exclusion criteria were enrolled and randomized to either Welchol 3.75 g (high-dose) or Welchol 0.625 g (low-dose).
Pre-assignment Details: Participants may have either been receiving metformin monotherapy or untreated with antidiabetic agents. All participants entered a 2-week, single-blind lead in/stabilization period after eligibility was confirmed. Metformin dose remained the same during the stabilization period.
Groups:
- Welchol 3.75 g (High-dose): Participants who were randomized to receive Welchol 3.75 g (high-dose) suspended in a drink for oral administration once daily with dinner.
- Welchol 0.625 g (Low-dose): Participants who were randomized to receive Welchol 0.625 g (low-dose) suspended in a drink for oral administration once daily with dinner.
Period: Overall Study
Arm/Group | Welchol 3.75 g (High-dose) | Welchol 0.625 g (Low-dose)
Started | 141 | 95
Completed | 99 | 72
Not Completed | 42 | 23
Not completed — Adverse Event | 8 | 3
Not completed — Lost to Follow-up | 11 | 6
Not completed — Withdrawal by Subject | 10 | 7
Not completed — Hyperglycemia meeting protocol-specified discontinuation criteria | 1 | 2
Not completed — Other | 12 | 5

BASELINE CHARACTERISTICS:
Population: Baseline demographic characteristics were assessed in the Randomized Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Welchol 3.75 g (High-dose) | Welchol 0.625 g (Low-dose) | Total
Number analyzed (Participants) | 141 | 95 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (2.09) | 14.2 (2.02) | 14.2 (2.06)
Age, Customized [Count of Participants; unit: Participants]
  10-13 years | 51 | 33 | 84
  14-17 years | 90 | 62 | 152
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 67 | 181
  Male | 27 | 28 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 49 | 38 | 87
  White | 71 | 46 | 117
  More than one race | 15 | 5 | 20
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 141 | 95 | 236

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Hemoglobin A1c (HbA1c) From Baseline to Month 6
Description: The percent change in HbA1c from baseline to Month 6 was assessed with the last observation after 1 month before any rescue therapy carried forward.
Time Frame: Baseline to Month 6 post-dose
Population: Change in HbA1c levels were assessed in the Intent-to-Treat population.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Welchol 3.75 g (High-dose) | Welchol 0.625 g (Low-dose)
Number analyzed (Participants) | 132 | 88
percent change | 0.09 [-0.18 to 0.36] | 0.21 [-0.11 to 0.54]
Statistical Analysis 1: Comparison: Welchol 3.75 g (High-dose) vs Welchol 0.625 g (Low-dose); Test type: Superiority; p = 0.5494, ANCOVA; Based on a mixed effect ANCOVA model with treatment and previous type 2 diabetes treatment stratum as fixed effects and baseline as a covariate; LS mean difference = -0.13, 95% CI 2-sided [-0.54 to 0.29], Standard Error of Mean 0.210

2. Secondary Outcome: Percent Change in Hemoglobin A1c (HbA1c) From Baseline to Month 12
Description: as for outcome 1
Time Frame: Baseline to Month 12 post-dose
Population: Change in HbA1c levels were assessed in the Intent-to-Treat population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Welchol 3.75 g (High-dose) | Welchol 0.625 g (Low-dose)
Number analyzed (Participants) | 122 | 83
percent change
  Month 3 | -0.27 [-0.49 to -0.06] | -0.05 [-0.31 to 0.22]
  Month 6: number analyzed (Participants) | 93 | 62
  Month 6 | -0.12 [-0.38 to 0.14] | -0.06 [-0.37 to 0.26]
  Month 9: number analyzed (Participants) | 65 | 38
  Month 9 | -0.06 [-0.42 to 0.30] | -0.16 [-0.61 to 0.30]
  Month 12: number analyzed (Participants) | 52 | 32
  Month 12 | -0.31 [-0.61 to -0.01] | -0.38 [-0.76 to 0.01]
  Month 12/Early termination: number analyzed (Participants) | 70 | 40
  Month 12/Early termination | -0.19 [-0.54 to 0.15] | -0.10 [-0.55 to 0.35]

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Month 12
Description: Change from baseline was assessed for FPG values at Month 6 and Month 12 categorical time points.
Time Frame: Baseline to Month 12 post-dose
Population: FPG values were assessed in the Intent-to-Treat population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Welchol 3.75 g (High-dose) | Welchol 0.625 g (Low-dose)
Number analyzed (Participants) | 90 | 61
mg/dL
  Month 6 | 11.6 [1.8 to 21.4] | 16.7 [4.7 to 28.7]
  Month 12: number analyzed (Participants) | 44 | 27
  Month 12 | 15.5 [2.9 to 28.1] | 10.6 [-5.8 to 27.0]
  Month 12/Early termination: number analyzed (Participants) | 50 | 27
  Month 12/Early termination | 14.6 [2.9 to 26.4] | 11.6 [-4.5 to 27.7]

4. Secondary Outcome: Number of Participants Achieving a Response to Therapy to Month 12
Description: Participants achieving a response to therapy, ie, glycemic control, were assessed with the last observation after 1 month before any rescue therapy carried forward at Month 6 and Month 12. Response to therapy was defined as HbA1c <7.0% or <6.5%, reduction in HbA1c ≥0.7% or ≥0.5% from baseline, and/or reduction in FPG ≥30 mg/dL from baseline.
Time Frame: Baseline to Month 12 post-dose
Population: Response to therapy was assessed in the Intent-to-Treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Welchol 3.75 g (High-dose) | Welchol 0.625 g (Low-dose)
Number analyzed (Participants) | 132 | 88
Participants
  Month 6 (LOCF): Achieving HBA1C <7% | 39 | 26
  Month 6 (LOCF): Achieving HBA1C <6.5% | 26 | 11
  Month 6 (LOCF): Achieving a reduction in HBA1C of ≥0.7% | 32 | 20
  Month 6 (LOCF): Achieving a reduction in HBA1C of ≥0.5% | 44 | 32
  Month 6 (LOCF): Achieving a reduction in FPG ≥30 mg/dL | 17 | 10
  Reduction in HBA1C of ≥0.7% and/or in FPG of ≥30 mg/dL from baseline to Month 6 with & without LOCF | 37 | 25
  Reduction in HBA1C of ≥0.5% and/or in FPG of ≥30 mg/dL from baseline to Month 6 with & without LOCF | 49 | 36
  Month 12: Achieving HBA1C <7% | 26 | 18
  Month 12: Achieving HBA1C <6.5% | 19 | 8
  Month 12: Achieving a reduction in HBA1C of ≥0.7% | 15 | 11
  Month 12: Achieving a reduction in HBA1C of ≥0.5% | 19 | 16
  Month 12: Achieving a reduction in FPG ≥30 mg/dL | 4 | 0
  Reduction in HBA1C of ≥0.7% and/or in FPG of ≥30 mg/dL from baseline to Month 12 | 15 | 11
  Reduction in HBA1C of ≥0.5% and/or in FPG of ≥30 mg/dL from baseline to Month 12 | 19 | 16
  Month 12/Early termination: Achieving HBA1C <7% | 33 | 19
  Month 12/Early termination: Achieving HBA1C <6.5% | 21 | 8
  Month 12/Early termination: Achieving a reduction in HBA1C of ≥0.7% | 20 | 13
  Month 12/Early termination: Achieving a reduction in HBA1C of ≥0.5% | 27 | 18
  Month 12/Early termination: Achieving a reduction in FPG ≥30 mg/dL | 5 | 0
  Reduction in HBA1C of ≥0.7% and/or in FPG of ≥30 mg/dL from baseline to Month 12/Early termination | 21 | 13
  Reduction in HBA1C of ≥0.5% and/or in FPG of ≥30 mg/dL from baseline to Month 12/Early termination | 28 | 18

5. Secondary Outcome: Percent Change From Baseline to Month 6 in Plasma Lipids
Description: The percent change in plasma lipids from baseline to Month 6 was assessed with the last observation after 1 month before any rescue therapy carried forward.
Time Frame: Baseline to Month 6 post-dose
Population: Change in lipid values were assessed in the Intent-to-Treat population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Welchol 3.75 g (High-dose) | Welchol 0.625 g (Low-dose)
Number analyzed (Participants) | 117 | 77
percent change
  Total cholesterol | 1.0 [-1.3 to 3.4] | 3.2 [0.3 to 6.1]
  Low-density lipoprotein cholesterol: number analyzed (Participants) | 115 | 76
  Low-density lipoprotein cholesterol | -1.1 [-4.7 to 2.4] | 4.4 [0 to 8.8]
  High-density lipoprotein cholesterol | 1.9 [-0.8 to 4.7] | 2.3 [-1.1 to 5.7]
  Non-High-density lipoprotein cholesterol | 1.2 [-1.9 to 4.2] | 4.1 [0.4 to 7.8]
  Apolipoprotein A-1 | 2.3 [0.2 to 4.5] | 3.1 [0.4 to 5.7]
  Apolipoprotein B | 0.8 [-2.0 to 3.5] | 2.7 [-0.7 to 6.2]

6. Secondary Outcome: Percent Change From Baseline to Month 6 in Triglycerides
Description: The percent change in triglycerides from baseline to Month 6 was assessed with the last observation after 1 month before any rescue therapy carried forward.
Time Frame: Baseline to Month 6 post-dose
Population: Triglyceride values were assessed in the Intent-to-Treat population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Welchol 3.75 g (High-dose) | Welchol 0.625 g (Low-dose)
Number analyzed (Participants) | 117 | 77
mg/dL | 10.0 [2.8 to 17.8] | 6.4 [-3.8 to 15.8]

7. Secondary Outcome: Number of Participants Requiring Rescue Medication Who Initially Met Rescue Criteria
Description: Rescue criteria was defined as HbA1c levels ≥8.5% after 3 months or ≥7.5% after 6 months (≥173 days) (confirmed persistent hyperglycemia) of study medication treatment, as measured by the central laboratory.
Time Frame: Baseline to Month 12 post-dose
Population: Participants meeting rescue criteria were assessed in the Intent-to-Treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Welchol 3.75 g (High-dose) | Welchol 0.625 g (Low-dose)
Number analyzed (Participants) | 132 | 88
Participants
  Met rescue criteria 1 time | 16 | 8
  Took rescue medication after meeting criteria 1 time | 4 | 0
  Did not take rescue medication after meeting criteria 1 time | 12 | 8
  Met rescue criteria 2 times | 18 | 5
  Took rescue medication after meeting criteria 2 times | 12 | 3
  Did not take rescue medication after meeting criteria 2 times | 6 | 2
  Met rescue criteria >2 times | 50 | 45
  Took rescue medication after meeting criteria >2 times | 43 | 42
  Did not take rescue medication after meeting criteria >2 times | 7 | 3
  Initially met rescue criteria at Month 3 to <Month 6 | 25 | 19
  Initially met rescue criteria at Month 6 to <Month 9 | 41 | 29
  Initially met rescue criteria at Month 9 to <Month 12 | 9 | 6
  Initially met rescue criteria at >Month 12 | 9 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were assessed from the date the participant signs the informed consent form up to the end of the study assessment and follow-up period, up to approximately 58 weeks.
Arm/Group | Welchol 3.75 g (High-dose) | Welchol 0.625 g (Low-dose)
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/95
Serious Adverse Events (participants affected / at risk) | 10/141 | 9/95
Other Adverse Events (participants affected / at risk) | 85/141 | 51/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Welchol 3.75 g (High-dose) (N=141) | Welchol 0.625 g (Low-dose) (N=95)
Affective disorder (Psychiatric disorders) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Premature labor (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abnormal behavior (Psychiatric disorders) | 0 | 1
Conversion disorder (Psychiatric disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Welchol 3.75 g (High-dose) (N=141) | Welchol 0.625 g (Low-dose) (N=95)
Abdominal pain (Gastrointestinal disorders) | 8 | 4
Abdominal pain upper (Gastrointestinal disorders) | 12 | 9
Constipation (Gastrointestinal disorders) | 10 | 1
Diarrhea (Gastrointestinal disorders) | 13 | 10
Nausea (Gastrointestinal disorders) | 8 | 7
Vomiting (Gastrointestinal disorders) | 20 | 11
Pyrexia (General disorders) | 7 | 5
Upper respiratory tract infection (Infections and infestations) | 24 | 9
Urinary tract infection (Infections and infestations) | 7 | 6
Joint sprain (Injury, poisoning and procedural complications) | 3 | 6
Nasopharyngitis (Infections and infestations) | 10 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 18 | 14
Headache (Nervous system disorders) | 17 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-08-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT01258075/Prot_SAP_000.pdf